CLINICAL TRIAL: NCT00759681
Title: A Prospective, Multi-center, Randomized Study to Evaluate the Safety and Efficacy of ArterX Vascular Sealant.
Brief Title: ArterX Surgical Sealant, A Randomized Prospective Multicenter Trial
Acronym: StEPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tenaxis Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLN-004; IDE Number - G070211
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2013-01-31 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2012-12

CONDITIONS: Vascular Disease
Keywords: Arterial Surgery; Open vascular Surgery; Sealant
MeSH Terms: conditions — Vascular Diseases | interventions — Gelatin Sponge, Absorbable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Gelfoam and Thrombin
  Interventions: Device: Gelfoam and Thrombin
- Investigational Device (Experimental): ArterX Surgical Sealant
  Interventions: Device: ArterX Surgical Sealant

INTERVENTIONS:
Device: ArterX Surgical Sealant — Apply at the suture site.
  Other Names: ArterX Vascular Sealant
  Arms: Investigational Device
Device: Gelfoam and Thrombin — Apply at the suture site.
  Other Names: Gelfoam Plus
  Arms: Control

SUMMARY:
This is a prospective, multi-center randomized, controlled study. The study is designed to assess the safety effectiveness of the ArterX Vascular Sealant compared to the control group in the open surgical repair of large vessels using synthetic vascular grafts or patches.

DETAILED DESCRIPTION:
To evaluate, during open vascular surgery, the safety and effectiveness of the ArterX™ Vascular Sealant when applied prophylactically. Application will be at synthetic vascular graft or patch to native vessel anastomosis prior to the restoration of full systemic circulation to achieve suture line sealing.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following criteria to be eligible for treatment in the Study:

1. The subject must be equal or greater than 18 years old.
2. The subject must be scheduled for the surgical placement of a synthetic (i.e., PTFE/Dacron) vascular graft or patch for large vessel repair/arterial reconstruction/hemodialysis access/arteriotomy.
3. The subject has no child bearing potential or has a negative serum or urine pregnancy test within 7 days of the index procedure.
4. The subject is willing and able to be contacted for the follow up visits at 6 weeks (± 7 days) and 3 months (± 7 days).
5. The subject or guardian must provide written informed consent using a form that is reviewed and approved by the IRB.

Exclusion Criteria:

Subjects will be excluded from the Study if any of the following criteria are met:

1. The subject has a known hypersensitivity or contraindication to heparin, bovine or seafood products.
2. The subject has a history of bleeding diathesis or coagulopathy, or will refuse blood transfusions.
3. The subject is currently enrolled in this, or another investigational device or drug trial (IDE or IND) that has not completed the required follow-up period. Note: Extended follow-up trials for products that were investigational but are currently commercially available are not considered investigational trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Cull, MD, Principal Investigator — Greenville Hospital System
Locations (1):
- Greenville Memorial Hospital, Greenville, South Carolina, United States

REFERENCES:
- [Result] Stone WM, Cull DL, Money SR. A randomized prospective multicenter trial of a novel vascular sealant. Ann Vasc Surg. 2012 Nov;26(8):1077-84. doi: 10.1016/j.avsg.2012.02.013. Epub 2012 Aug 29. PMID 22939276

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 217 subjects (110 ArterX, 107 Control) were treated at eleven (11) participating investigational centers. Randomized subjects were treated from 10/08 to 12/09. The last follow-up visit was conducted in 03/10.
Groups:
- Control: Gelfoam and Thrombin: Gelfoam PlusTM is used to seal suture lines of arterial grafts or patches made from PTFE and Dacron. Gelfoam is a sterile compressed sponge and Thrombin is the last enzyme in the clotting cascade.
- Investigational Device: ArterX Surgical Sealant: ArterX is a two-component sealant provided in a double barreled syringe. The main components are bovine serum albumin and a polyaldehyde formed from polymerized glutaraldehyde. The solutions are dispensed through a double plunger, mixing the two components in a 1:1 ratio by passing them through a specially designed mixing tip, delivering up to 2 ml volume of each component.
Period: Overall Study
Arm/Group | Control: Gelfoam and Thrombin | Investigational Device: ArterX Surgical Sealant
Started | 107 | 110
Completed | 97 | 100
Not Completed | 10 | 10
Not completed — Death | 2 | 5
Not completed — Lost to Follow-up | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Control: Control Treatment: Gelfoam and Thrombin
- Investigational Device: Investigational Treatment: ArterX Surgical Sealant
- Total: Total of all reporting groups
Arm/Group | Control | Investigational Device | Total
Number analyzed (Participants) | 107 | 110 | 217
Age Continuous [Mean (Standard Deviation); unit: years] | 65.7 (12.3) | 66.2 (12.3) | 66.0 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 41 | 78
  Male | 70 | 69 | 139
Region of Enrollment [Number; unit: participants]
  United States | 107 | 110 | 217

OUTCOME MEASURES:

1. Primary Outcome: Immediate Sealing Evidenced by no Bleeding on Clamp Release.
Description: The immediate sealing evidenced by no bleeding on clamp release was measured at time of surgery
Time Frame: Immediate at time of surgery
Population: Treatment sites were the unit of measure based on ITT for effectiveness outcomes.
Measure: Number; unit: Treatment sites
Units Other Than Participants: Treatment sites
Groups:
- Control Treatment: Control Treatment: Gelfoam and Thrombin
- Investigational Device: Investigational Device: ArterX Surgical Sealant
Arm/Group | Control Treatment | Investigational Device
Number analyzed (Participants) | 107 | 110
Number analyzed (Treatment sites) | 164 | 167
Treatment sites | 65 | 101
Statistical Analysis 1: Comparison: Control Treatment vs Investigational Device; Effectiveness was evaluated using a superiority hypothesis, comparing treatment sites with regards to the proportion achieving immediate suture line sealing between the groups. Effectiveness was based on a two-tailed, 0.05 hypothesis test, with a minimum effect size set at 10%. The mean difference in the proportion of sites achieving immediate suture line sealing was compared between the Control and Investigation Device groups; Test type: Superiority or Other; p = 0.05, Exact binomial confidence limit; Effectiveness: 95% confidence limits of the difference between groups, and ensuring that the lower limit of the difference was greater than 10%; Mean Difference (Final Values) = 0.208, 95% CI 2-sided [0.103 to 0.314], Standard Error of Mean 0.0538

2. Primary Outcome: Cumulative Incidence of Significant Bleeding, Infection, Neurological Deficit or Inflammatory/Immune Allergic Response
Description: The Primary Safety Endpoint Will be the Cumulative Incidence of Significant Bleeding, Infection, Neurological Deficit or Inflammatory/Immune Allergic Response Through 6 Weeks.
Time Frame: Treatment through 6 weeks
Population: Based on ITT population for primary safety analysis.
Measure: Number; unit: participants
Groups:
- Control Treatment: Control Treatment with Gelfoam and Thrombin
Arm/Group | Control Treatment | Investigational Device
Number analyzed (Participants) | 107 | 110
participants | 64 | 51
Statistical Analysis 1: Comparison: Control Treatment vs Investigational Device; The mean difference is equivalent to the proportion of Investigational Device patients minus the proportion of Control patients experiencing any instance of significant bleeding, neurological deficit or immune/inflammatory allergic response; Test type: Non-Inferiority or Equivalence — Safety was evaluated using non-inferiority hypothesis evaluating the proportion of cases with any instance of sign. bleeding, neurological deficit or immune/inflammatory allergic response. Safety based on one-tailed, 0.05 alpha, with equivalence limit set at 15%; p = 0.05, Exact binomial confidence limit; Safety: 95% confidence limits of the difference between groups, and ensuring that the upper limit of the difference was less than or equal to 15%; Mean Difference (Final Values) = -0.135, 95% CI 1-sided [upper limit -0.003], Standard Error of Mean 0.0671 — The cumulative incidence of safety endpoints for the Investigational Treatment group was an average of 13.5% less than for the Control group

ADVERSE EVENTS:
Time Frame: Adverse events were collected through 3 months post surgery.
Description: Adverse events were collected from surgery through hospital discharge, and at each follow-up visit, 6 weeks and 3 months post-surgery.
Groups:
- 2. Gelfoam and Thrombin: Gelfoam and Thrombin
- 1. ArterX Surgical Sealant: ArterX Surgical Sealant
Arm/Group | 2. Gelfoam and Thrombin | 1. ArterX Surgical Sealant
Serious Adverse Events (participants affected / at risk) | 26/107 | 28/110
Other Adverse Events (participants affected / at risk) | 11/106 | 9/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 2. Gelfoam and Thrombin (N=107) | 1. ArterX Surgical Sealant (N=110)
Significant Bleeding (Surgical and medical procedures) | 2 | 3
Infection (Infections and infestations) | 19/106 | 9/108
Neurological Deficit (Nervous system disorders) | 2/105 | 3/108
Immune/Inflammatory Allergic Response (Immune system disorders) | 0/106 | 0/108
Death (Investigations) | 2 | 5
Hypotension (Vascular disorders) | 0 | 3
Thrombosis/Thromboembolism (Vascular disorders) | 1 | 3
Ischemia (Vascular disorders) | 1 | 2
Respiratory Failure/Dysfunction (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Steal Syndrome (Vascular disorders) | 0 | 2
Myocardial Infarction (Cardiac disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2. Gelfoam and Thrombin (N=106) | 1. ArterX Surgical Sealant (N=108)
Non-serious Infections (Infections and infestations) | 11 | 9 — For Other Adverse Events/non-serious infections, the denominator for the Control and Investigational groups are less than the total subjects at risk since 3 total subjects were not evaluated for non-serious infections since due to early termination.

LIMITATIONS AND CAVEATS:
There were no significant trial limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No